CLINICAL TRIAL: NCT04644783
Title: A Novel Blood Test to Predict Safe (Non-trigger) Foods for Infants and Toddlers With Food Protein-induced Enterocolitis Syndrome (FPIES)
Brief Title: Novel Blood Test to Predict Safe Foods for Infants and Toddlers With Food Protein-induced Enterocolitis Syndrome (FPIES)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Mohamad El-Zaatari, Research Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00156027
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Food Protein-Induced Enterocolitis Syndrome; Allergies; Pediatric Disorder
Keywords: Safe foods; Trigger foods; Vomiting
MeSH Terms: conditions — Hypersensitivity; Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Blood test with assays (Experimental): 10 participants with FPIES exhibiting reactions to more than 2 foods will be recruited.
  Interventions: Diagnostic Test: Blood test assay

INTERVENTIONS:
Diagnostic Test: Blood test assay — Participants will have their blood drawn and be evaluated with a new blood assay that screens a large number of foods (more than 20) in a culture plate. Participants will be asked to eat the identified safe foods by the the blood assay.

SUMMARY:
The aim of this study is to validate a blood test that can identify safe foods for food protein-induced enterocolitis syndrome (FPIES). This study proposes a solution to the problems of FPIES by developing a new blood assay that screens a large number of foods (more than 20) in a culture plate. If this blood test is successful it may be able to identify safe foods more quickly.

The study will recruit 10 participants that will have more than 2 trigger foods.

DETAILED DESCRIPTION:
Participants will complete surveys and have blood draws during the study. Additionally, participants will be asked to keep track of their diet as well as introduce safe foods identified by the researchers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FPIES
* Have to have documented reactions to 2-3 trigger foods with recurrent delayed vomiting or documented reactions to 4 or more trigger foods with recurrent delayed vomiting.

Exclusion Criteria:

* Patients who are currently on medications that suppress the immune system
* Patients who do not have at least 2 trigger foods identified.
* Patients who have a history of an organic Gastrointestinal (GI) disease (e.g., inflammatory bowel disease, celiac disease, biliary disorders, bowel resection), cardiac, pulmonary, neurologic, renal, endocrine, or gynecological pathology
* Lack of parental or guardian informed consent.

Ages: 1 Month to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad El Zaatari, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sanders GM, Hua A, Hudson E, Troost JP, Kamada N, Kao JY, Schuler CF 4th, El-Zaatari M. Association of myeloid cell reactivity patterns with safe food predictions in FPIES patients. Allergy Asthma Clin Immunol. 2025 May 21;21(1):24. doi: 10.1186/s13223-025-00968-1. PMID 40400028

RESULTS

PARTICIPANT FLOW:
Groups:
- Blood Test With Assays: 10 participants with FPIES exhibiting reactions to more than 2 foods were recruited.
  Blood test assay: Participants had their blood drawn and evaluated with a new blood assay that screened a large number of foods (more than 20) in a culture plate. Participants were asked to eat the foods identified as safe by the blood assay.
Period: Overall Study
Arm/Group | Blood Test With Assays
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Blood Test With Assays: 10 participants with FPIES exhibiting reactions to more than 2 foods were recruited.
  Blood test assay: Participants had their blood drawn and evaluated with a new blood assay that screened a large number of foods (more than 20) in a culture plate. Participants were asked to eat the foods identified as safe by the the blood assay.
Arm/Group | Blood Test With Assays
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 0.75 [0.5 to 2.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Negative Predictive Value (NPV), Defined as the Percentage of Test-predicted Safe Foods That Are Actually Safe Foods.
Description: A Receiver operating characteristic (ROC) curve was built to estimate the NPV. A random-effects logit model was used to model the binary outcome (safe or trigger food) as a function of the 9 biomarker measurements in the assay. (Expression Value = Relative fold change of 9-gene expression panel in response to food treatment, divided by fold change in response to LPS treatment, multiplied by 1000). The random effect in the logit model took into consideration the correlated data measured within the same subject. A cluster ROC curve analysis was used to assess the precision of the assay. Specifically, the area was computed under the cluster ROC curve (AUC). A threshold to obtain the NPV was selected based on inspection of the ROC curve.
  At the initial visit, participants had their blood drawn, which was assayed. On average, participants came in up to 4 weeks later after the test results were ready. Participants were then asked to trial a new food each week for up to 7 weeks.
Time Frame: Up to 7 weeks from the first blood trial, on average 11 weeks
Measure: Number; unit: percentage
Arm/Group | Blood Test With Assays
Number analyzed (Participants) | 10
percentage
  NPV <29.24 Threshold | 98.5
  Area Under the ROC Curve | 73.16
Statistical Analysis 1: Comparison: Blood Test With Assays; Test type: Superiority; p < 0.0001, Regression, non-linear mixed effects

2. Secondary Outcome: Positive Predictive Value (PPV), Defined as the Percentage of Test-predicted Unsafe Foods That Are Actually Unsafe Foods.
Description: The same ROC curve described for the primary outcome was used to derive the PPV. At the initial visit, participants had their blood drawn, which was assayed. On average, participants came in up to 4 weeks later after the test results were ready. Participants were then asked to trial a new food each week for up to 7 weeks.
Time Frame: Up to 7 weeks from the first blood trial, on average 11 weeks
Measure: Number; unit: percentage
Arm/Group | Blood Test With Assays
Number analyzed (Participants) | 10
percentage | 31.1
Statistical Analysis 1: Comparison: Blood Test With Assays; Test type: Superiority; p < 0.0001, Regression, non-linear mixed effects

ADVERSE EVENTS:
Time Frame: 4 months (after assay results were communicated)
Arm/Group | Blood Test With Assays
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT04644783/Prot_SAP_000.pdf